CLINICAL TRIAL: NCT03514368
Title: Monitoring of Immunological Mechanisms and Biomarkers Underlying Efficacy and Toxicity of Cancer Immunotherapy
Acronym: MINER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17 GENE 23
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Solid Cancers
Keywords: Immune checkpoint modulation; Tumor antigens; Adaptive immune responses; Tumor molecular signature
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients treated with immune checkpoint blockade (Other)
  Interventions: Other: Patients treated with immune checkpoint blockade

INTERVENTIONS:
Other: Patients treated with immune checkpoint blockade — Tumor biopsy specimens and blood samples will be collected at different time points:
  * Baseline
  * before the 3rd ICB administration (blood samples only)
  * before the 5th ICB administration (blood samples only)
  * at the time of treatment permanent discontinuation (blood samples only)
  * at the time of progression (tumor biopsy specimens only)
  * after the last dose of ICB treatment (blood samples only taken twice per year until study termination)

SUMMARY:
This trial is a translational, open-label, multi-site, prospective cohort study of 520 patients aiming to identify and to monitor immunological biomarkers associated with therapeutic response to immune checkpoints blockade (ICB), in patients with multiple types of advanced (unresectable and/or metastatic) solid cancers.

The study will be conducted on a population of patients receiving ICB (anti-PD-1 or anti-PD-L1 or anti-CTLA4, alone or in combination) in the context of either routine care or a clinical study protocol.

Patients with any of the following tumor types may be enrolled in the trial:

* Non-Small Cell Lung Cancer (NSCLC),
* Head and neck cancer,
* Melanoma,
* Bladder cancer,
* Other tumor types when Immuno-Oncology agent is expected to be efficient or when a clinical trial is an option.

For each included patient, tumor biopsy specimens and blood samples will be collected at different time points.

All included patients will be followed-up until progression. After this date, survival data will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of study entry.
2. Patient with histologically documented metastatic and/or unresectable solid malignant tumor (NSCLC, head and neck, melanoma (except uveal melanoma), bladder cancer or any other advanced solid tumor when I-O agent is expected to be efficient or when a clinical trial is an option).
3. Patient for which a treatment with immune checkpoint blockade including, but not limited to, anti-PD-1, anti-PD-L1 and anti-CTLA-4 mAb alone or in combination has been decided.
4. Archived tumor specimen available or feasible for pre-treatment tumor biopsy.
5. Current treatment with ICB not yet started.
6. Evaluable disease (measurable as per RECIST 1.1. or not).
7. ECOG Performance status 0-2.
8. Patient able to participate and willing to give informed consent prior to performance of any study-related procedures.
9. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Patient pregnant, or breast-feeding.
2. Uveal melanoma
3. Any condition contraindicated with tumor /blood sampling procedures required by the protocol.
4. Known history of positive test for hepatitis B virus or hepatitis C virus or human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
5. Any current severe or uncontrolled disease, including, but not limited to ongoing or active infection and auto immune disorders.
6. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
7. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Rate of objective response (complete or partial response) | 18 months by patient
  Response will be assessed according to RECIST 1.1 / investigator judgment

SECONDARY OUTCOMES:
Progression Free Survival defined as the time from inclusion until progression according to investigator judgment, or death, whichever occurs first. | 18 months by patient
Anti-tumor immune responses under immunotherapy defined by investigator judgment and/or iRECIST criteria | 18 months by patient
Immune related adverse event (irAE) will be evaluated using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 | 12 months by patient

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hopital Larrey, Toulouse
  - Institut Universitaire Du Cancer de Toulouse - Oncopole, Toulouse
  - Chu Rangueil, Toulouse